CLINICAL TRIAL: NCT03543891
Title: Correlation Study of Thyroid Cancer and Intestinal Microbiota
Brief Title: Intestinal Microbiota and Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2018-05-20
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2017-09

CONDITIONS: Microbiota
Keywords: Gut microbiota; 16S rRNA gene; Thyroid cancer; Metabonomics
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: 50 healthy volunteers were included in the healthy control group
- Thyroid cancer group: 50 patients of thyroid cancer were included

INTERVENTIONS:
Other:
  Groups: Thyroid cancer group

SUMMARY:
Thyroid cancer (TC), the most common malignancy of the endocrine system, is currently the fifth most common malignancy diagnosed in women (1). The incidence of TC in the United States has increased by an average of 3% per year over the past 4 decades. Much progress has been made in exploring the etiology and pathogenesis of thyroid cancer, while the exact etiology remains unknown, TC is thought to arise from interactions between genetic susceptibility factors, epigenetic effects, and various environmental factors. Besides the improvement of diagnosis, TC increasing incidence emphasize that other important factors such as the environment play an important role in disease pathogenesis. While microbiota as an environment factor to some cancers accept widespread attention, if microbiota also as a risk factor for TC, it is worthy to be considered.

DETAILED DESCRIPTION:
Thyroid cancer (TC), the most common malignancy of the endocrine system, is currently the fifth most common malignancy diagnosed in women (1). The incidence of TC in the United States has increased by an average of 3% per year over the past 4 decades. According to the China National Cancer Registry data in 2015 (3), there were estimated 90,000 new TC cases in China, and its incidence has risen sharply. Much progress has been made in exploring the etiology and pathogenesis of thyroid cancer, while the exact etiology remains unknown, TC is thought to arise from interactions between genetic susceptibility factors, epigenetic effects, and various environmental factors. Besides the improvement of diagnosis, TC increasing incidence emphasize that other important factors such as the environment play an important role in disease pathogenesis. While microbiota as an environment factor to some cancers accept widespread attention, if microbiota also as a risk factor for TC, it is worthy to be considered.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Patients of thyroid cancer

Exclusion Criteria:

* Pregnancy
* Lactation
* Cigarette smoking
* Alcohol addiction
* Hypertension
* Diabetes mellitus
* Lipid dysregulation
* BMI > 27
* Recent (< 3 months prior) use of antibiotics, probiotics, prebiotics, symbiotics, hormonal medication, laxatives, proton pump inhibitors, insulin sensitizers or Chinese herbal medicine
* History of disease with an autoimmune component, such as MS, rheumatoid arthritis, IBS, or IBD
* History of malignancy or any gastrointestinal tract surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients were included according to the inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Transcriptional changes in gut microbiota | Baseline
  The microbiota measured by 16S rRNA gene

SECONDARY OUTCOMES:
Metabolic changes in gut microbiota | Baseline
  Metabolic changes measured by metabonomics analysis

CONTACTS AND LOCATIONS:
Overall Officials: Yunwei Wei, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No